CLINICAL TRIAL: NCT00594217
Title: Determining the Rapidity With Which Exogenous P Suppresses Daytime LH (GnRH) Pulse Frequency in Women During the Follicular Phase of the Menstrual Cycle
Brief Title: Determining How Quickly Progesterone Slows LH Pulse Frequency
Acronym: CRM001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Chris McCartney, Associate Professor of Medicine, University of Virginia
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 13368; R01HD058671 (NIH)
Record Dates: First submitted 2008-01-04; First posted 2008-01-15 (Estimated); Results first posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Normal; PCOS
Keywords: PCOS
MeSH Terms: interventions — Progesterone

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled, crossover study
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PCOS women (Experimental): PCOS women: women were considered to have PCOS if they had evidence of clinical and/or biochemical hyperandrogenism plus oligo-/amenorrhea in the absence of other identifiable causes.
  Interventions: Drug: oral micronized progesterone suspension; Other: Placebo
- Normal Controls (Active Comparator): Normal control women: women with regular menstrual cycles without evidence of hyperandrogenism.
  Interventions: Drug: oral micronized progesterone suspension; Other: Placebo

INTERVENTIONS:
Drug: oral micronized progesterone suspension — oral micronized progesterone suspension, single 100 mg oral dose
  Other Names: progesterone
Other: Placebo — Placebo contains only inert ingredients and is not expected to exert any direct physiological effects

SUMMARY:
The rapidity with which progesterone (P) suppresses daytime lutenizing hormone (LH) (and by inference gonadotropin releasing hormone (GnRH)) pulse frequency is unknown. We propose to assess this further using a randomized, cross-over, placebo-controlled study. Ovulatory women will begin E2 patches on day 4-8 of the cycle, while women with PCOS will begin E2 patches either on day 4-8 of the cycle or at least 8 weeks post-menses. After 3 d of E2 administration, women will undergo a 24-h sampling study in the GCRC. Beginning at 2000 h, blood for LH, FSH, E2, P, and T will be obtained over a 24-h period. After 10 h of sampling, either oral micronized P (100 mg p.o.) suspension or placebo suspension will be administered (according to randomization). At the completion of sampling, E2 patches will be discontinued. During a subsequent menstrual cycle (or after at least 3 weeks in oligomenorrheic PCOS), subjects will undergo another GCRC study identical to the first (including pretreatment with E2) except that oral P will be exchanged for placebo or vice versa in accordance with the crossover design. We will assess the acute effects of progesterone on LH frequency, with secondary endpoints being mean LH, LH pulse amplitude, and mean follicle-stimulating hormone (FSH). We propose two primary hypotheses: (1) administration of P (at 0600 h) to normally cycling adult women during the follicular phase will result in a demonstrable suppression of daytime LH (and by inference GnRH) pulse frequency within 12 hours; (2) administration of P (at 0600 h) to women with PCOS will result in less suppression of daytime LH pulse frequency than in ovulatory women without PCOS. A secondary hypothesis is that augmentation of LH amplitude after P administration will be less in PCOS compared to normal controls.

DETAILED DESCRIPTION:
Studies under this protocol will be performed in normally cycling women and in women with PCOS from 18 to 35 years old. Criteria for PCOS will be (a) clinical and/or biochemical evidence of hyperandrogenism, (b) oligomenorrhea, and (b) the absence of clinical or biochemical evidence of other potential causes of hyperandrogenism and/or oligomenorrhea. After informed consent is obtained, all potential subjects will undergo a screening history and physical exam. Subjects will need to fast for a minimum of 8 hours prior to screening blood draw. After informed consent is obtained, blood tests (~ 16 cc) will be drawn at 0800-0900 h as follows: LH, FSH, progesterone (P), estradiol (E2), total testosterone, SHBG, 17-OHP, androstenedione, DHEA-S, beta-hCG, TSH, prolactin, CBC, chemistry and liver panels, hemoglobin A1c, fasting insulin, and fasting glucose. Additionally, BOD POD® will be used to measure total fat mass, fat free mass, and percent body fat. Waist and hip circumference will be measured.

This study follows a crossover design, with assessment of the acute effects of P and placebo (individually) on GnRH pulse frequency; subjects will be randomized to receive either P or placebo during the first GCRC admission, with subsequent GCRC study occurring during a subsequent cycle.

Women will begin E2 patches (0.1 mg/d per patch, 2 patches [delivering a total of 0.2 mg/d] placed on the abdomen and changed every 2 d) on the evening of day 4-8 of the study cycle (controls or PCOS) or >= 8 weeks post-menses (PCOS only). These patches will be continued for a total of 4 d, with GCRC admission occurring on day 3 of E2 administration. Exogenous E2 administration will standardize hypothalamic exposure to E2 and help ensure the presence of sufficient hypothalamic P receptors.

Four to 5 days before a scheduled GCRC admission, subjects will come to the GCRC for an outpatient blood draw for P and beta-HCG (2 cc). If 30 days will have elapsed between (a) the most recent hemoglobin and hematocrit and (b) the scheduled GCRC admission, a hemoglobin and hematocrit will also be drawn at this time (1cc).

After 3 d of E2 administration, women will undergo a 24-h sampling study in the GCRC. Estradiol administration (E2 patches) will continue throughout the GCRC admission. Subjects will be admitted to the GCRC at 1800 h (2 h prior to sampling). Beginning at 2000 h, blood will be obtained through an indwelling i.v. forearm heparin lock over a 24-h period as follows: LH every 10 min (1 ml); P every 30 min (1 ml); FSH, E2, and T every 2 h (assays to be run in same samples as LH and P). SHBG, fasting insulin, and fasting glucose (i.e., fasting since 2200 h) will be run on the 0600 h sample (extra 2 cc drawn). (Subjects will fast from 2200 to 0600 h.) After 10 h of sampling (i.e., at 0600 h), either oral micronized P (100 mg p.o.) suspension or placebo suspension will be administered (according to randomization). With exogenous P, we aim to achieve mean plasma P concentrations 4-8 ng/ml. Subjects will not be allowed to sleep during the day (i.e., from 0600 to 2200 h). Subjects will be encouraged to sleep from 2200 to 0600. Sleep will be formally evaluated (extraoculograms, electroencephalograms, wrist actigraphy, etc.). At the completion of sampling, E2 patches will be discontinued. Volunteers will be discharged on oral iron (325 mg BID). We will ask women to eat only the food provided by the GCRC.

Subjects will undergo another GCRC study identical to the first (including pretreatment with E2, outpatient blood draw 4-5 days before admission, etc.), except that oral P will be exchanged for placebo or vice versa in accordance with the crossover design. (Subjects will again begin E2 patches on the evening of cycle day 4-8 [controls or PCOS] or >= 8 weeks post-menses [PCOS only].) In this way, we will be able to standardize any change in GnRH pulse frequency after P administration to any change in GnRH pulse frequency after placebo administration.

The study will end after the second GCRC admission. Subjects will be asked to continue oral iron supplementation for at least 30 d after this last GCRC admission.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be healthy women in two groups: (1) women with regular menstrual cycles and no evidence of hyperandrogenism, and (2) women with PCOS (defined as clinical/biochemical evidence of hyperandrogenism plus oligomenorrhea, but with no evidence for other endocrinopathies).
* Subjects will be 18-35 years old.
* Subjects will be willing to strictly avoid pregnancy (using non-hormonal methods) during the time of study and must be willing and able to provide informed consent.

Exclusion Criteria:

* We will exclude women with a history of any disorders that may potentially be complicated by hormonal treatment, such as DVT and breast, ovarian, or endometrial cancer.
* We will exclude women with any other cancer diagnosis and/or treatment (with the exception of basal cell or squamous skin carcinoma) unless they have remained clinically disease free (based on appropriate surveillance) for five years.
* Women with anemia (hematocrit < 36% and/or a hemoglobin level <12 g/dl) will be treated with iron for a maximum of 2 sequential months before the 1st admission and/or before the 2nd admission. If they remain anemic after 2 sequential months of ferrous gluconate (325 mg bid), they will then be excluded from further participation in the study.
* Women with a history of any disorders that may potentially be complicated by long-term iron supplementation, such as hemochromatosis and polycythemia vera, will be excluded.
* Women with a significant history of cardiac or pulmonary dysfunction (e.g., known or suspected congestive heart failure; known or suspected coronary atherosclerosis; asthma requiring systemic intermittent corticosteroids; etc.) will be excluded.
* Women with liver enzymes, alkaline phosphatase, or bilirubin > 1.5 times upper limit of normal (confirmed on repeat) will be excluded, with the exception that mild bilirubin elevations will be accepted in the setting of known Gilbert's syndrome.
* Abnormal sodium or potassium concentrations (confirmed on repeat); bicarbonate concentrations <20 or >30 (confirmed on repeat)
* Women with abnormal renal function (i.e., serum creatinine > 1.4) will be excluded (confirmed on repeat)
* Pregnant and breast-feeding women will be excluded.
* A history of allergy to progesterone or estradiol will constitute grounds for exclusion.
* Women with a BMI greater or equal to 40 kg/m2.
* Virilization
* A total testosterone > 150 ng/dl in women with PCOS (which suggests the possibility of a virilizing neoplasm) (confirmed on repeat)
* Elevated DHEAS (mild elevations may be seen in PCOS, and elevations < 1.5 times the upper limit of normal will be accepted in PCOS) (confirmed on repeat)
* Follicular 17-hydroxyprogesterone > 300 ng/dl, which suggests the possibility of congenital adrenal hyperplasia (if elevated during the luteal phase and there is a concern about the possibility of congenital adrenal hyperplasia, the 17-hydroxyprogesterone may be collected during the follicular phase, or >60 if oligomenorrheic). NOTE: If a 17-hydroxyprogesterone > 300 ng/dl is confirmed on repeat testing, an ACTH stimulated 17-hydroxyprogesterone < 1000 ng/dl will be required for study participation.
* A previous diagnosis of diabetes, a fasting glucose ≥ 126 mg/dl, or a hemoglobin A1c > 6.5%
* Abnormal TSH (subjects with adequately treated hypothyroidism, reflected by normal TSH values, will not be excluded; or, for a new diagnosis of hypothyroidism, further study will at the least be delayed pending appropriate treatment) (confirmed on repeat)
* Abnormal prolactin (mild elevations may be seen in PCOS, and elevations < 1.5 times the upper limit of normal will be accepted in this group) (confirmed on repeat)
* Evidence of Cushing's syndrome by history or physical exam
* Due to the amount of blood being drawn in the study, subjects with body weight < 110 lbs. will be excluded from the study

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 85 (Actual)
Dates: Start 2007-11-29 (Actual); Primary Completion 2020-01-18 (Actual); Study Completion 2020-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher McCartney, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided
We do not have current plans to share IPD

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 85 subjects enrolled in this study. 29 women initiated formal study procedures. However, for personal reasons, 4 women dropped out of the study after completing only 1 admission. In addition, data from one woman was excluded from analysis because her study was unintentionally performed during the luteal phase. Thus, data for 24 women were formally analyzed. 56 women were withdrawn from study prior to being assigned to an arm of intervention.
Groups:
- PCOS Women: PCOS women: women were considered to have PCOS if they had evidence of clinical and/or biochemical hyperandrogenism plus oligo-amenorrhea in the absence of other identifiable causes.
- Normal Controls: Normal controls: non-PCOS women with regular menstrual cycles and without evidence of hyperandrogenism.
Period: Overall Study
Arm/Group | PCOS Women | Normal Controls
Started | 13 | 16
Completed | 12 | 13
Not Completed | 1 | 3
Not completed — Withdrawal by Subject | 1 | 3

BASELINE CHARACTERISTICS:
Population: Data from one woman in the control group was excluded from analysis because her average progesterone level before progesterone administration was 4.8 ng/mL (15.3 nmol/L), indicating that the frequent-sampling study was unintentionally performed during the luteal phase.
Groups:
- Total: Total of all reporting groups
Arm/Group | PCOS Women | Normal Controls | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants] — Ages 18 - 35 years
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 12 | 12 | 24
    >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 4 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 9 | 7 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: LH Pulse Frequency
Description: The primary endpoint is the change in the number of LH pulses (over 10 hours) attributable to progesterone.
Time Frame: 10 hours before and after administration of micronized progesterone and placebo
Measure: Median (Inter-Quartile Range); unit: pulses/hour
Arm/Group | PCOS Women | Normal Controls
Number analyzed (Participants) | 12 | 12
pulses/hour
  Placebo 20:00-06:00 (pre-pbo) | 1.31 [1.01 to 1.88] | 0.91 [0.81 to 1.44]
  Placebo 10:00-20:00 (post-pbo) | 1.33 [1.24 to 1.85] | 1.19 [1.04 to 1.52]
  Progesterone 20:00-06:00 (pre-P4) | 0.99 [0.80 to 1.85] | 0.98 [0.86 to 1.44]
  Progesterone 10:00-20:00 (post-P4) | 1.18 [.97 to 1.76] | 1.05 [1.01 to 1.44]

2. Secondary Outcome: Mean LH
Description: A secondary endpoint is the change in mean LH concentration (over 10 hours) attributable to progesterone.
Time Frame: 10 hours before and after administration of micronized progesterone and placebo
Measure: Median (Inter-Quartile Range); unit: IU/L
Arm/Group | PCOS Women | Normal Controls
Number analyzed (Participants) | 12 | 12
IU/L
  Placebo 20:00-06:00 (pre-pbo) | 8.2 [7.8 to 34.4] | 6.4 [3.9 to 10.3]
  Placebo 10:00-20:00 (post-pbo) | 12.0 [9.6 to 36.0] | 8.8 [7.1 to 16.5]
  Progesterone 20:00-06:00 (pre-P4) | 8.6 [7.6 to 18.1] | 5.6 [2.5 to 17.6]
  Progesterone 10:00-20:00 (post-P4) | 26.6 [20.9 to 50.0] | 20.7 [10.6 to 54.9]

3. Secondary Outcome: LH Pulse Mass
Description: A secondary endpoint is the change in LH pulse mass (a correlate of LH pulse amplitude) attributable to progesterone.
Time Frame: 10 hours before and after administration of micronized progesterone and placebo
Measure: Median (Inter-Quartile Range); unit: IU/L
Arm/Group | PCOS Women | Normal Controls
Number analyzed (Participants) | 12 | 12
IU/L
  Placebo 20:00-06:00 (pre-pbo) | 3.6 [2.5 to 6.7] | 4.85 [4.0 to 13.6]
  Placebo 10:00-20:00 (post-pbo) | 4.3 [2.9 to 8.2] | 7.51 [5.3 to 26.4]
  Progesterone 20:00-06:00 (pre-p4) | 3.6 [1.7 to 11.1] | 5.47 [3.8 to 15.8]
  Progesterone 10:00-20:00 (post-p4) | 13.9 [7.5 to 32.2] | 13.96 [9.3 to 35.4]

4. Secondary Outcome: Mean FSH
Description: A secondary endpoint is the change in mean FSH concentration (over 10 hours) attributable to progesterone.
Time Frame: 10 hours before and after administration of micronized progesterone and placebo
Measure: Median (Inter-Quartile Range); unit: IU/L
Arm/Group | PCOS Women | Normal Controls
Number analyzed (Participants) | 12 | 12
IU/L
  Placebo 20:00-06:00 (pre-pbo) | 4.5 [3.0 to 6.3] | 3.5 [3.1 to 5.4]
  Placebo 10:00-20:00 (post-pbo) | 3.9 [3.3 to 9.0] | 4.5 [3.8 to 7.0]
  Progesterone 20:00-06:00 (pre-p4) | 4.2 [3.0 to 6.4] | 4.4 [2.5 to 5.9]
  Progesterone 10:00-20:00 (post-p4) | 6.3 [4.4 to 9.1] | 8.0 [5.63 to 14.6]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected beginning after subjects began study drug/intervention/study-related procedures/specimen collection up until the end of the study drug/intervention/participation; an average of 6 months.
Arm/Group | PCOS Women | Normal Controls
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/16
Other Adverse Events (participants affected / at risk) | 3/13 | 3/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PCOS Women (N=13) | Normal Controls (N=16)
nausea (Gastrointestinal disorders) | 1 | 0
Spotting (Reproductive system and breast disorders) | 0 | 2
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 | 0
fatigue (General disorders) | 1 | 0
swelling at IV site (Skin and subcutaneous tissue disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Results of this study have been published and are publicly available at https://pmc.ncbi.nlm.nih.gov/articles/PMC8981178/

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-04-11): https://cdn.clinicaltrials.gov/large-docs/17/NCT00594217/Prot_SAP_001.pdf
  • Informed Consent Form (2017-05-16): https://cdn.clinicaltrials.gov/large-docs/17/NCT00594217/ICF_000.pdf